CLINICAL TRIAL: NCT04610736
Title: TEMOkids Study: A Population Pharmacokinetic, Acceptability and Safety Study for KIMOZO, a Paediatric Oral Suspension of Temozolomide
Brief Title: TEMOkids Study : A Phase I Pediatric Study for KIMOZO, Oral Suspension of Temozolomide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orphelia Pharma (Industry)
Collaborators: ClinSearch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORP-TMZ-I- b
Record Dates: First submitted 2020-10-20; First posted 2020-10-30 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Cancer
Keywords: neuroblastoma; other pediatric cancers requiring temozolomide
MeSH Terms: conditions — Neoplasms; Neuroblastoma

STUDY DESIGN:
Intervention Model Description: Non-randomized, international, multi-centre, open-label, single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Temozolomide 40 mg/ml, Oral suspension
  Interventions: Drug: Temozolomide Oral Suspension

INTERVENTIONS:
Drug: Temozolomide Oral Suspension — One prescribed oral dose (range 75 to 200 mg/m2) once daily for 5 days
  Other Names: KIMOZO, Ped-TMZ

SUMMARY:
Non-randomized, international, multi-centre, open-label, single arm study to determine the pharmacokinetic (PK) parameters of a single dose of an oral suspension of temozolomide (KIMOZO) in the pediatric population aged 1 year and over.

DETAILED DESCRIPTION:
The TEMOkids study is an international open-label, non-randomized, prospective, single-arm phase 1 study to determine the pharmacokinetic (PK) parameters of a single dose of an oral suspension of temozolomide (KIMOZO) in the pediatric population aged 1 year and over.

Patients will be subject to at least one 21 or 28-day treatment cycle involving administration of an oral suspension of temozolomide (KIMOZO) for five consecutive days followed by 16 or 23-days resting period, with determination of the PK parameters on the first treatment day.

Five (5) additional cycles will be allowed under compassionate use regimen. The compassionate use period could be extended at the discretion of the investigator and in agreement with the sponsor. Safety and activity data will be collected during the compassionate follow-up period.

The study will be held in multiple sites spread across Europe.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients in need of temozolomide (all indications with 5-day treatment per 21- or 28-day cycle).
* Male and female patients aged 1 to less than 18 years
* Patients who have signed the informed consent or for which one, both parents or legal guardian (depending on local legislation) have signed the informed consent.
* Patients having records of coverage by a health insurance
* Life expectancy ≥ 3 months
* Adequate haematological function:

  * haemoglobin ≥ 80 g/L (transfusion support authorized)
  * neutrophil count ≥ 1.0 x 10e9 cells/L
  * platelet count ≥ 100 x 10e9 cells/L (without transfusion support)
  * in case of bone marrow involvement: neutrophils ≥ 0.5 x 10e9 cells/L and platelets ≥75 x 10e9 cells/L
* Adequate renal function:

  * Creatine clearance ≥ 60 mL/min.1.73m² according to the Schwartz formula [1] or its modified form [2]
* Adequate hepatic function:

  * bilirubin ≤1.5 x ULN
  * AST and ALT ≤ 2.5 x ULN (AST, ALT 5xULN in case of liver metastases)
* Lansky Score ≥ 70%

Exclusion Criteria:

* Patients who are co-administrated at day one with sodium valproate as it decreases the clearance of temozolomide
* Patients with (naso)gastric tube administration of temozolomide during first cycle of treatment.
* Patients already enrolled in studies investigating temozolomide or other investigational new drugs.
* A post-menarche female with a positive blood/urine pregnancy test at inclusion.
* Known contraindication or hypersensitivity to temozolomide or any chemically close substance

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Population Phamacokinetic parameter: AUC24 | At Day 1 of treatment cycle 1 (each cycle is 21 or 28 days) with post-dose samples collected at about 0.15, 0.5, 1, 2.5, and 7 hours post dose
  Estimated by a population analysis performed with NONMEM (7.4)
Population Phamacokinetic parameter: Cmax | At Day 1 of treatment cycle 1 (each cycle is 21 or 28 days) with post-dose samples collected at about 0.15, 0.5, 1, 2.5, and 7 hours post dose
  Estimated by a population analysis performed with NONMEM (7.4)
Population Phamacokinetic parameter: T1/2 | At Day 1 of treatment cycle 1 (each cycle is 21 or 28 days) with post-dose samples collected at about 0.15, 0.5, 1, 2.5, and 7 hours post dose
  Estimated by a population analysis performed with NONMEM (7.4)

SECONDARY OUTCOMES:
Acceptability of the oral suspension of temozolomide: score | At Day 1 and Day 5 of treatment cycle 1 (each cycle is 21 or 28 days)
  Scoring with a standardized assessment tool: CAST - ClinSearch Acceptability Score Test®. This tool measures 9 observational drivers of drug acceptability.
Incidence of treatment-emergent adverse events | Through study completion, an average of 6 months including compassionate use period
  Adverse events collected directly by investigators when patient is hospitalized and through patient diary completed by caregivers and medically controlled by investigators when patient is at home
Activity of the oral suspension of temozolomide | At the end of each 21- or 28-day treatment cycle of the compassionate use period
  Activity assessment (complete or partial response, stable disease, disease progression)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Abbou, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (11):
- France (5):
  - Centre Oscar Lambret, Lille
  - Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon
  - CHU Timone Enfants, Marseille
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif
- Germany (2):
  - Charité University Medicine Berlin, Berlin
  - Hopp Children's Cancer Center Heidelberg, Heidelberg
- Princess Maxima Center for Pediatric Oncology, Utrecht, Netherlands
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No